CLINICAL TRIAL: NCT00797901
Title: Depression Treatment in General Medical Settings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Puerto Rico (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Mildred Vera, Ph.D., University of Puerto Rico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S06GM008224 (NIH)
Record Dates: First submitted 2008-11-24; First posted 2008-11-25 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Collaborative Care, Treatment as Usual (Experimental)
  Interventions: Other: Collaborative Care

INTERVENTIONS:
Other: Collaborative Care

SUMMARY:
The purpose of this study was to examine the effect of a new disease management model for depression, the Collaborative Depression Management Program (CDMP), designed to improve clinical outcomes and increase depression treatment in general medical settings.

DETAILED DESCRIPTION:
Clinically depressed individuals that could benefit from newer treatments for depression often do not receive care. Low treatment rates are of particular concern since depression is projected to be the second leading cause of disability worldwide by 2010. Major depression has been the focus of numerous intervention studies with primary care patients during recent years. However, despite advances in the development and testing of quality intervention models for depression treatment, very little is known about the effectiveness of interventions with Latinos. This is important because Latinos are less likely than whites to receive depression treatment, even though the rates of depression are similar for both groups. A major public health challenge is to make available the benefits of intervention developments in depression treatment for all groups in society. As a first step, we examined the impact of a quality depression intervention with Puerto Ricans. The specific aims were:

1. To examine the effect of a Collaborative Depression Management Program in reducing depressive symptoms, improving quality of life, and decreasing health-related functional impairment among Puerto Rican patients in general medical settings.
2. To determine whether a Collaborative Depression Management Program is effective in improving satisfaction with care and reducing barriers to depression treatment among Puerto Rican patients in general medical settings.

This study employed a randomized experimental design. Depressed patients receiving general medical care were assigned to one of two conditions: 80 to the Depression Management Program and 80 to treatment as usual. All subjects completed assessments at baseline, week 8, week 16 and week 24. Our overall programmatic goals were to increase the likelihood that depressed patients receive care and to make available for the Puerto Rican community advances in the treatment of major depression.

ELIGIBILITY:
Inclusion Criteria:

* patients ages 18 or older that meet the clinical criteria for major depression.

Exclusion Criteria:

* pregnancy, planning a pregnancy, breastfeeding or less than 3 months post-partum
* severe cognitive impairment
* ongoing psychiatric treatment
* do not plan to use the study clinic as a main source of medical care during the next six months
* a history of bipolar disorder or psychosis
* those clinically judged to have a high acute suicidal risk
* unstable or life-threatening medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2004-08; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Depression | 2 months
Health-Related Functional Impairment | 2 months
Quality of Life | 2 months

SECONDARY OUTCOMES:
Satisfaction with Care | 2 months
Barriers to Treatment | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Mildred Vera, Ph.D., Principal Investigator — University of Puerto Rico; Deborah Juarbe, Ph.D., Study Director — University of Puerto Rico
Locations (1):
- University of Puerto Rico, San Juan, Puerto Rico